CLINICAL TRIAL: NCT03938441
Title: Biweekly Interval Intermittent Fasting for Type 2 Diabetes, a Safety Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment and PI Graduating Residency in June 2021.
Sponsor: gino gaddini (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, gino gaddini, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWH20190059H
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Type 2; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent Fasting (Experimental): Modified 5:2 intermittent fasting
  Interventions: Other: Intermittent Fasting

INTERVENTIONS:
Other: Intermittent Fasting — The version of 5:2 intermittent fasting to be applied in this study will be somewhat less intensive than implemented then what has been proposed in some recent, similar studies.
  On fasting days, instead of limiting the subject to a specific calorie count, the subject will be instead instructed to skip either the first or last meal of the day in order to complete a 12 to 16 hour fast, during which time they are allowed drink water or any non-caloric beverage of their choice, but not consume any calories.
  Furthermore, the patient will be instructed for their remaining 2 meals to consume no more than they would on a normal, non-fasting day.

SUMMARY:
The purpose of this study is to establish safety of biweekly intermittent fasting in the setting of type 2 diabetes mellitus or prediabetes under treatment with non-hypoglycemic agents (e.g. metformin).

DETAILED DESCRIPTION:
This study is proposed as a prospective interventional cohort safety study for biweekly intermittent fasting.

In the effort to improve compliance of lifetime dietary change, the version of 5:2 intermittent fasting to be applied in this study will be somewhat less intensive than implemented then what has been proposed in some recent, similar studies.

On fasting days, instead of limiting the subject to a specific calorie count, the subject will be instead instructed to skip either the first or last meal of the day in order to complete a 12 to 16 hour fast, during which time they are allowed drink water or any non-caloric beverage of their choice, but not consume any calories.

Furthermore, the patient will be instructed for their remaining 2 meals to consume no more than they would on a normal, non-fasting day.

ELIGIBILITY:
**Subjects must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and female Active Duty members and DoD beneficiaries ages 18-69
* Diagnosed with Type 2 Diabetes or pre-diabetic
* Prescribed/taking Metformin 500mg to 2000mg daily

Exclusion Criteria:

* History of recurrent hypoglycemic events on present medication regimen
* Drugs/medication with known increase in hypoglycemic events [Include basal insulin, rapid acting insulin, sulfonylureas, etc.). Metformin is not known to cause hypoglycemia.
* Pregnant
* Medication-induced or secondary diabetes
* Known abnormal hematocrit

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic events | Number will vary depending on the number of hypoglycaemic events per each subject and will be recorded throughout study until completion at 12 weeks
  This study's intent is to investigate the safety of this intervention for use in a broader scope. It is imperative that risks are known for each subpopulation of diabetics. To this point, our literature review indicates that hypoglycemic events did occur at higher rates in fasting populations taking hypoglycemic medications. We intend to look at rates of hypoglycemia on those not on hypoglycemic medications to assess if this trend continues.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Study Director — US Air Force
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Carter S, Clifton PM, Keogh JB. The effects of intermittent compared to continuous energy restriction on glycaemic control in type 2 diabetes; a pragmatic pilot trial. Diabetes Res Clin Pract. 2016 Dec;122:106-112. doi: 10.1016/j.diabres.2016.10.010. Epub 2016 Oct 19. PMID 27833048
- [Background] Arnason TG, Bowen MW, Mansell KD. Effects of intermittent fasting on health markers in those with type 2 diabetes: A pilot study. World J Diabetes. 2017 Apr 15;8(4):154-164. doi: 10.4239/wjd.v8.i4.154. PMID 28465792
- [Background] Azevedo FR, Ikeoka D, Caramelli B. Effects of intermittent fasting on metabolism in men. Rev Assoc Med Bras (1992). 2013 Mar-Apr;59(2):167-73. doi: 10.1016/j.ramb.2012.09.003. PMID 23582559
- [Background] Ash S, Reeves MM, Yeo S, Morrison G, Carey D, Capra S. Effect of intensive dietetic interventions on weight and glycaemic control in overweight men with Type II diabetes: a randomised trial. Int J Obes Relat Metab Disord. 2003 Jul;27(7):797-802. doi: 10.1038/sj.ijo.0802295. PMID 12821964
- [Background] Horne BD, Muhlestein JB, Anderson JL. Health effects of intermittent fasting: hormesis or harm? A systematic review. Am J Clin Nutr. 2015 Aug;102(2):464-70. doi: 10.3945/ajcn.115.109553. Epub 2015 Jul 1. PMID 26135345
- [Background] Corley BT, Carroll RW, Hall RM, Weatherall M, Parry-Strong A, Krebs JD. Intermittent fasting in Type 2 diabetes mellitus and the risk of hypoglycaemia: a randomized controlled trial. Diabet Med. 2018 May;35(5):588-594. doi: 10.1111/dme.13595. Epub 2018 Feb 27. PMID 29405359
- [Background] Genuth S, Eastman R, Kahn R, Klein R, Lachin J, Lebovitz H, Nathan D, Vinicor F; American Diabetes Association. Implications of the United kingdom prospective diabetes study. Diabetes Care. 2003 Jan;26 Suppl 1:S28-32. doi: 10.2337/diacare.26.2007.s28. No abstract available. PMID 12502617
- [Background] Centers for Disease Control and Prevention. National Diabetes Statistics Report, 2017. Atlanta, GA: Centers for Disease Control and Prevention, U.S. Dept of Health and Human Services; 2015.